CLINICAL TRIAL: NCT01138865
Title: Effect of Continuous Positive Airway Pressure (CPAP) on Cardiovascular Biomarkers in Patients With Obstructive Sleep Apnea.
Brief Title: Effect of CPAP on Biomarkers in Patients With OSA
Acronym: CPAP
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, S.K.SHARMA, Professor and Haed, All India Institute of Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SKS/CPAP-OSAS/2009
Record Dates: First submitted 2010-06-02; First posted 2010-06-08 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive sleep apnea; Cytokine levels; Insulin resistance; Hypertension; Dyslipidemia; Albumin-creatinine ratio; Continuous positive airway pressure (CPAP)
MeSH Terms: conditions — Sleep Apnea, Obstructive; Insulin Resistance; Hypertension; Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other): Device: AutoSet Spirit--Wash--Modified-AutoSet Spirit 3 months of therapeutic CPAP (auto-titrating CPAP) followed by 3 months of non-therapeutic sham-CPAP with 1 month of wash-out in between
  Interventions: Device: AutoSet Spirit--Wash--Modified-AutoSet Spirit
- 2 (Other): 3 months of non-therapeutic sham-CPAP followed by 3 months of therapeutic CPAP (auto-titrating CPAP) with 1 month of wash-out in between
  Interventions: Device: Modified-AutoSet Spirit--Wash-AutoSet Spirit

INTERVENTIONS:
Device: AutoSet Spirit--Wash--Modified-AutoSet Spirit — 3 months of therapeutic CPAP (auto-titrating CPAP) followed by 3 months of non-therapeutic sham-CPAP with 1 month of wash-out in between
  Other Names: AutoSet Spirit(TM), ResMed India Ltd.
  Arms: 1
Device: Modified-AutoSet Spirit--Wash-AutoSet Spirit — 3 months of non-therapeutic sham-CPAP followed by 3 months of therapeutic CPAP (auto-titrating CPAP) with 1 month of wash-out in between
  Other Names: Modified-AutoSet Spirit(TM), ResMed India Ltd.
  Arms: 2

SUMMARY:
CPAP, the standard treatment for Obstructive sleep apnea syndrome (OSAS) that reduces sleep fragmentations and neurocognitive deficit in OSAS may also have a key role in reduction of cardiovascular, mortality risks in the same patients.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a condition in which there is collapse of the upper airway during sleep, as a result of which there is a decrease or complete cessation of airflow. This leads to repeated episodes of hypoxia during sleep and sleep fragmentation. It is a highly prevalent though under-recognized clinical problem.There is increasing evidence that inflammation plays important role in development of cardiovascular complications in patients with OSA.

Continuous positive airway pressure (CPAP) is the standard treatment for OSA with significant symptoms.However, it is a costly treatment option and poor compliance is an important limiting factor. CPAP treatment has been shown to improve the daytime somnolence and neurocognitive function in people with OSAS. However, its effect on cardiovascular biomarkers in people with OSAS has not been satisfactorily assessed.

This study aims to assess the effect of CPAP treatment on cardiovascular biomarkers in OSA.

ELIGIBILITY:
Inclusion Criteria:

The 1st part of the study will include

1. males and females, aged 30-65 years,
2. with AHI >5 and excessive daytime sleepiness
3. naïve to CPAP treatment.
4. Subjects from first part of the study who have moderately severe OSAS and have never received treatment for OSA,diabetes mellitus and hypertension

Exclusion Criteria:

1. Hypothyroidism
2. Chronic renal failure
3. Chronic liver disease
4. Chronic lung disease
5. Known systemic inflammatory diseases (lupus , sarcoidosis and other connective tissue disorders),
6. Use of drugs that influence urinary protein excretion (eg. steroids, lithium, NSAIDS, ACE inhibitors/Angiotensin Receptor Blockers etc.)
7. Immune deficiency conditions
8. Pregnancy
9. Active menstruation at time of sampling
10. Macroalbuminuria (aACR>300mg/g),
11. Patients of coronary artery disease and left ventricular dysfunction
12. Not on treatment for hypertension, diabetes mellitus or dyslipidemia
13. Long lasting hypertension or diabetes mellitus (more than 5 years after diagnosis)

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-03; Primary Completion 2014-09 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Effect of CPAP therapy on blood pressure | 7 months
Effect of CPAP therapy on insulin resistance | 7months
Effect of CPAP therapy on plasma hs-CRP | 7months
Effect of CPAP therapy on lipid profile | 7months
Effect of CPAP therapy on urinary albumin-creatinine ratio | 7months

SECONDARY OUTCOMES:
Effect of CPAP on anthropometric parameters | 3 months
Effect of CPAP on visceral fat and other imagings | 3months
Effect of CPAP on carotid intima medical thickness | 3months
Effect of CPAP on adipokines and oxidative stress markers | 3months
Effect of CPAP on inflammatory cytokine levels. | 3months

CONTACTS AND LOCATIONS:
Overall Officials: Surendra K Sharma, MD,Ph.D, Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India